CLINICAL TRIAL: NCT03082040
Title: Effects of a Home-based Breathing Training on Menopausal Symptoms Among Community Menopausal Women
Brief Title: A Home-based Breathing Training on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yuh-Kae Shyu, Assistant Professor, Ministry of Science and Technology, Taiwan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOST105-2314-B-030-006
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Menopause; Menopause Related Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will undergo a home-based breathing training 20 minutes twice daily for four weeks
  Interventions: Behavioral: home-based breathing training
- waiting-list control group (Other): Participants in the control condition will conduct the same breathing training as the intervention group after a four-week waiting list period
  Interventions: Behavioral: home-based breathing training

INTERVENTIONS:
Behavioral: home-based breathing training — The intervention group will undergo a home-based breathing training 20 minutes twice daily for four weeks. Participants in the control condition will participate the same breathing training after a four-week waiting list period.

SUMMARY:
This is a prospective, triple-blinded and randomized controlled trial examining the effects of a home-based breathing training assisted with biofeedback on menopausal symptoms and autonomic functions among community menopausal women. We also examines whether the changes in autonomic functions would be mediators between slow breathing and menopausal symptoms. This study will include menopausal women, aged from 45 to 64, who experienced menopausal symptoms. Participants will be randomly assigned to either an intervention group (n = 80) or a waiting-list control group (n = 80). The intervention group will undergo the home-based breathing training 20 minutes twice daily and participants in the control condition will participate the same breathing training after a four-week waiting list period. The primary outcome measures are menopausal symptoms measured by symptom diaries of menopausal symptoms and the Greene Climacteric Scale (GCS). Secondary outcome measures are autonomic functions expressed by blood pressure (BP), heart rate (HR) and heart rate variability (HRV). Measurements will be taken at baseline, week 4, and week 8.

DETAILED DESCRIPTION:
Ditto

ELIGIBILITY:
Inclusion Criteria:

* aged from 45 to 64, reporting cessation of menstrual cycles with natural causes ≧ 12 consecutive months
* the Greene Climacteric Scale (GCS) Chinese version scores ≧ 1

Exclusion Criteria:

* clinically diagnosed with history of cardiac arrhythmia, coronary heart disease, heart failure, kidney disease, hypertension, chronic low blood pressure, diabetic neuropathy, psychosis or mental deficiency
* received hormone replacement therapy prescribed by gynecological physicians
* took cardiac medications which may affect the autonomic functions, ex., β-blockers, etc.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Menopausal symptoms | Baseline
  Assessments using the Greene Climacteric Scale (GCS) for self-reported menopausal symptoms
Menopausal symptoms | Posttest (4 weeks from baseline)
  Assessments using the Greene Climacteric Scale (GCS) for self-reported menopausal symptoms

SECONDARY OUTCOMES:
Autonomic functions (Blood pressure) | Baseline
  Assessments using A&D sphygmomanometer (Model 767Plus, A&D Co., LTD., Japan) for systolic blood pressure and diastolic blood pressure
Autonomic functions (Blood pressure) | Posttest (4 weeks from baseline)
  Assessments using A&D sphygmomanometer (Model 767Plus, A&D Co., LTD., Japan) for systolic blood pressure and diastolic blood pressure
Autonomic functions (heart rate) | Baseline
  Assessments using EKG sensors to detect heartbeat signals, and then be analyzed by the BioGraph Infiniti software.
Autonomic functions (heart rate) | Posttest (4 weeks from baseline)
  Assessments using EKG sensors to detect heartbeat signals, and then be analyzed by the BioGraph Infiniti software.
Autonomic functions (heart rate variability) | Baseline
  A 3-lead EKG and Cardiopro Software were used to assess and analyze the heart rate variability in time domain, including SDNN (standard deviation of all NN intervals), rMSSD (the root mean square successive difference of normal-to-normal intervals) and pNN50 (NN50 count divided by the total number of all NN intervals).
Autonomic functions (heart rate variability) | Posttest (4 weeks from baseline)
  A 3-lead EKG and Cardiopro Software were used to assess and analyze the heart rate variability in time domain, including SDNN (standard deviation of all NN intervals), rMSSD (the root mean square successive difference of normal-to-normal intervals) and pNN50 (NN50 count divided by the total number of all NN intervals).

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Kae Shyu, PhD, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University, New Taipei City, Xinzhuang Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No